CLINICAL TRIAL: NCT05692661
Title: A Dose Escalation Study of Proton and Carbon Ion Irradiation for HER2 Positive and Triple Negative Breast Cancer After Breast Conserving Surgery
Brief Title: A Dose Escalation Study of Proton and Carbon Ion Irradiation for HER2 Positive and Triple Negative Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Qing Zhang,MD, Professor, Shanghai Proton and Heavy Ion Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-BCa2022-01
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Triple Negative Breast Cancer; HER2-positive Breast Cancer
Keywords: Breast Cancer; HER2 Positive; Triple Negative; Proton and Carbon Ion; Dose Escalation
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — Protons; Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- proton plus carbon ion radiotherapy (Experimental): CTV1: whole breast, proton therapy. CTVboost: Tumor bed, carbon ion dose escalation study with four dose levels.
  Interventions: Radiation: proton plus carbon ion radiotherapy

INTERVENTIONS:
Radiation: proton plus carbon ion radiotherapy — CTV1: whole breast, 40.05Gy(RBE) in 15 fractions with proton ion therapy; CTVboost: Tumor bed, carbon ion dose escalation study with four dose levels [10.2Gy(RBE)/3Fx,10.8Gy(RBE) /3Fx,11.4Gy(RBE)/3Fx and 12Gy(RBE)/3Fx ].

SUMMARY:
Adjuvant radiotherapy is the standard treatment for early breast cancer after breast conserving surgery. Molecular subtypes was significantly associated with the risk of local recurrence of breast cancer. Nguyen et al found that the overall 5-year cumulative incidence of local recurrence was 0.8% for luminal A, 1.5% for luminal B, 8.4% for HER2 positive, and 7.1% for triple negative breast cancer after lumpectomy and radiotherapy. Her2 positive and triple negative breast cancers may be inherently radioresistant.

Therefore, for HER2 positive and triple negative breast cancer with high local recurrence and radiation resistance, proton combined with carbon ion is proposed after breast conserving surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HER2 positive or Triple Negative invasive breast carcinoma.(HER2 positive: immunohistochemistry [IHC] 3+ and or fluorescence in situ hybridization [FISH] amplified; Triple Negative: estrogen receptor [ER] and progesterone receptor [PR] < 1%, HER2 negative [IHC 1+ or 2+ FISH non-amplified])
* Age ≥ 18 years and ≤ 80 years.
* The primary tumor must be excised via breast conserving surgery.
* Stage p T1-2 N0 M0
* ECOG performance status ≤2.

Exclusion Criteria:

* Invasive breast cancer not confirmed by pathology.
* Distant metastasis
* Prior thoracic radiation.
* Pregnancy or lactating.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-10 (Estimated); Primary Completion 2025-10-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | 3 months after the completion of CIRT
  Treatment related acute toxicity assessed by CTCAE v4.03

SECONDARY OUTCOMES:
Local regional recurrence | within 5 years after radiotherapy.
  The Ipsilateral breast and regional lymph nodes recurrence
Cosmetic outcome as measured by Breast Cancer Treatment Outcomes Scale | within 5 years after radiotherapy.
  Cosmetic outcome will be evaluated by Breast Cancer Treatment Outcomes Scale filled out by patients.
Cosmetic outcome as measured by BCCT.core software | within 5 years after radiotherapy.
  Patients' photographs of the breasts will be taken. With the use of BCCT.core software from The Breast Research group (INESC TEC) cosmetic outcome will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Proton and Heavy Ion center, Shanghai, China